CLINICAL TRIAL: NCT06434480
Title: Stereotactic Body Radiotherapy (SBRT) in Advanced Hepatocellular Carcinoma With Oligoprogression on Atezolizumab Plus Bevacizumab
Brief Title: SBRT in HCC With Oligoprogression on Atezo-Bev
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Landon Chan, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC078
Record Dates: First submitted 2024-05-14; First posted 2024-05-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: HCC
Keywords: SBRT in HCC
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Experimental): After screening procedures, suitable patients are consented and enrolled with the following treatment being given
  * Continue Atezolizumab 1200mg Day 1 plus Bevacizumab 15mg/kg Day 1, given intravenously every 3 weeks, till the next progression, or death.
  * Radiotherapy will start 4 to 6 weeks after consent
  * For intrahepatic progression: 27.5-50Gy in 5 fractions over 2 weeks will be given.
  * For extrahepatic progression: an aim to give ablative dose (i.e. BED10≥100Gy) will be given (allow lower dose based on nearby OAR dose constraints and is at the discretion of the treating radiation oncologist)
  * Bevacizumab will need to be withhold 4 weeks prior and after radiotherapy.
  * Dose constraints to organ at risk (OAR) will take reference from RTOG-1112 and UK 2022 consensus on normal tissue dose-volume constraints
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy (SBRT) — * For intrahepatic progression: 27.5-50Gy in 5 fractions over 2 weeks will be given.
  * For extrahepatic progression: an aim to give ablative dose will be given.

SUMMARY:
HCC is a huge healthcare burden in Hong Kong and is one of the top 5 cancers in terms of incidence and mortality in Hong Kong. Patients with advanced HCC are treated with immunotherapy-based combination atezolizumab plus bevacizumab as first-line treatment as a standard of care. At the moment, there is limited evidence to guide subsequent treatments after patients progressed on atezolizumab plus bevacizumab. Oligoprogression is a term used to describe patients who had limited progression (usually less than 3 sites) on systemic therapy, with the rest of the lesions controlled. Previous studies in non-HCCs have shown that addition of locoregional treatment (e.g. radiotherapy) may prolong the use of systemic therapy, resulting in improved survival, but this has been relatively unexplored for HCC. In this prospective, single-arm study, we aim to evaluate the treatment outcome, efficacy and safety of the addition of radiotherapy to oligoprogressive sites for patients who had limited progression on atezolizumab plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years old
2. ECOG performance 0 to 1
3. Confirmed diagnosis of HCC
4. Oligoprogression on Atezolizumab plus Bevacizumab, as defined as ≤3 lesions (intra- and extrahepatic lesions all together; vascular tumor thrombus is counted as one lesion)
5. Progressed lesion(s) amenable to SBRT:

   * At most one site of intrahepatic and one site of extrahepatic lesion will be irradiated
   * For intrahepatic progression:

     * Number of intrahepatic progression ≤ 3
     * Total intrahepatic tumours ≤ 5
     * Maximum sum of HCC ≤ 20cm
     * Any one HCC ≤ 15cm
     * Normal liver volume minus intrahepatic GTV > 700cc
     * Mean liver dose ≤ 15Gy
     * No measurable common or main branch biliary duct involvement
     * No direct tumor invasion into the stomach, duodenum, small bowel or large bowel
   * For extrahepatic progression:

     * Maximal tumor size ≤ 3cm
     * Respective dose constraints of organ at risks as listed on the UK 2022 Consensus on Normal Tissue Dose-Volume Constraints for Oligometastatic, Primary Lung and Hepatocellular Carcinoma Stereotactic Ablative Radiotherapy can be met.
6. Prior radiofrequency ablation (RFA) or trans-arterial chemoembolization (TACE) are eligible
7. Child-Pugh A liver function
8. Life expectancy longer than 12 weeks
9. At least one measurable treatment lesion according to RECIST 1.1
10. Written informed consent must be obtained prior to any study related procedures
11. Adequate haematological function (Hb ≥ 8.5g/dL; Plt ≥ 75x109/L; ANC ≥ 1.5x109/L; INR ≤ 1.5)
12. Adequate hepatic function (albumin ≥ 28g/l; Bilirubin ≤ 1.5xULN; ALT < 5 times upper limit normal)
13. Adequate renal function (serum creatinine ≤ 1.5 times the upper limit of normal range; Na ≥ 130mmol/L; K ≥ 3.0mmol/L)
14. Able to read, understand and provide written consent

Exclusion Criteria:

1. History of another malignancy except appropriately-treated BCC of skin or CIN of cervix during the last 5 years
2. Previous radiotherapy to the abdomen
3. Previous yttrium-90 chemoembolization
4. Repetitive history of non-healing wounds or ulcers within 2 months of inclusion
5. Pregnant or lactating females at any time during the study
6. Active autoimmune disease requiring systemic therapy in the past 2 years
7. Diagnosis of immunodeficiency (including HIV)
8. Ongoing corticosteroid therapy >10mg prednisone daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) with the addition of SBRT to oligo-progressive sites | 2 years

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
Objective response rates (ORR) of the irradiated lesion(s) | 2 years
Overall objective response rates (ORR) | 2 years
Additional treatment related adverse events (TRAE) | 2 years
Pattern of progression | 2 years
  Four types of progression pattern:
  * EHG (extrahepatic growth)
  * IHG (intrahepatic growth)
  * NEH (new extrahepatic lesion)
  * NIH (new intrahepatic growth)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No